CLINICAL TRIAL: NCT02015585
Title: Evaluation of Mandibular Movements and Condyle-fossa Relation From Two Treatment Protocols. A Randomized Clinical Trial.
Brief Title: Evaluation of Influence of Two Treatment Protocols on Mandibular Movements and Condyle-fossa Relation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Clinical Trials Coordinator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO0014
Record Dates: First submitted 2013-09-13; First posted 2013-12-19 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Interocclusal appliance (Experimental): Patients will be submitted to the treatment with interocclusal appliances 30 days before the replacement of their complete dentures.
  Interventions: Procedure: interocclusal appliance; Procedure: Complete denture rehabilitation
- Relining complete denture base (Experimental): Patients will be submitted to a procedure of relining their old dentures 30 days before the replacement of the complete dentures.
  Interventions: Procedure: Relining of the complete dentures; Procedure: Complete denture rehabilitation
- Only Rehabilitation (Active Comparator): Patients will be treated with a complete denture without any kind of previous intervention
  Interventions: Procedure: Complete denture rehabilitation

INTERVENTIONS:
Procedure: interocclusal appliance — Patients will be submitted to the treatment with interocclusal appliances 30 days before the replacement of their complete dentures.
  Arms: Interocclusal appliance
Procedure: Relining of the complete dentures — Patients will be submitted to the relining of their old dentures 30 days before the replacement of their complete dentures.
  Arms: Relining complete denture base
Procedure: Complete denture rehabilitation — All patients will be rehabilitated with new complete dentures in the study

SUMMARY:
The edentulism and use of inadequate dentures, unstable and with teeth worn because long period of usage can lead to an disharmony of the stomatognathic system due to gradual loss of occlusion vertical dimension resulting in inadequate mandibular movements and condyle-fossa relation. The reline of the denture base and the use of interocclusal appliance prior to definitive rehabilitation could have influence on these functional aspects. However, there are not Randomized Controlled clinical Trials (RCTs) testing the combined use of these two treatments in reestablishing these functional aspects. The, aim of this study is to evaluate whether the denture base reline and the use of interocclusal appliance prior to final rehabilitation have influence on mandibular movements and condyle-fossa relation, incomplete denture wearers. For this controlled, crossover, randomized and blinded clinical trial, 30 volunteers, totally edentulous, complete denture wearer over a period of five year, will be selected. The volunteers will be randomly allocated into three subgroups (n= 10) and will receive the following treatments: Control (C)Volunteers will receive new complete denture without any previous intervention in their old complete denture; Relining Denture (RD)Volunteers will be submitted to the relining of the base of the their old complete denture and after 30 days of usage and before the replacement of the new complete denture, an evaluation will be performed; Interocclusal Appliance (IA) Volunteers will be submitted to the treatment with interocclusal appliance and after 30 days of usage and before the replacement of the new complete denture, an evaluation will be performed. Volunteers will be evaluated regarding the extent of mandibular movement by intraoral record of Gothic Gysi arch; condyle-fossa relation by cone-bean computed tomographic scan; occlusion vertical dimension by Willis compass and photographic record. These evaluations will be performed at three periods, T0 baseline; T1 after application of randomized treatment, reline denture and interocclusal appliance); T3 after final rehabilitation. The control group will be evaluated only at periods T0 and T3.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults suffering from upper and lower denture indicated for replacement due to use exceeding five years;
2. Have availability to attend FO / UFPel days predetermined;
3. Agree with the term informed consent, approved by the research ethics committee of FO / UFPel.

Exclusion Criteria:

1. Patients younger than 40 years;
2. Patients who are not users of denture upper and lower;
3. Patients denture wearers during periods of less than five years.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the occlusal vertical dimension after treatment at 6 months | 30 days after randomization; and 30 days after final prosthetic rehabilitation

SECONDARY OUTCOMES:
Change from baseline in the extension of the mandibular movements up to 6 months. | 30 days after randomization; and 30 days after the final prosthetic rehabilitation
  The extent of mandibular movement will be assessed by intramural record of Gothic Gysi arch.

OTHER OUTCOMES:
Change from baseline in the condyle-fossa relation up to six months | 30 days after randomization; and 30 days after the final prosthetic rehabilitation
  The condyle-fossa relation will be measured by cone-bean computed tomographic scan.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil